CLINICAL TRIAL: NCT05103930
Title: Innovation for Participation
Brief Title: InnovationForParticipation
Acronym: I4P
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: InnovationForParticipation
Record Dates: First submitted 2021-08-10; First posted 2021-11-02 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Children; Disabilities
Keywords: assistive products; technology; children with disabilities; life situation

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Children with disabilities experience activities limitations and participation restrictions. Facilitating the children with disabilities' independence while performing tasks is a key stake to improve their successful participation and their development.

Products and technology can prevent, compensate, relieve or neutralize disability or handicap and help children and youth with disabilities to perform tasks that might otherwise be difficult or impossible.

The aim of this study was i) to identify the most frequent activity limitations and participation restrictions for which assistive products and technology may be useful for children and youth with disabilities, and ii) to highlight macroscopic trends related to encountered difficulties and wished products and technology.

The hypotheses were i/ that difficulties would be particularly expected for certain life situations, especially outside the home in an unfamiliar environment ii/ that products and technology would be wished for those situations which should be defined as priority subjects and iii/ that thanks to those results it could be possible to highlight new processes to develop innovative solutions.

DETAILED DESCRIPTION:
The study was conducted according to current French legislation (loi Jardé (n°2012-300).It was a cross-sectional study with a convergent parallel mixed method design. It used an online open survey following the STROBE and CHERRIES guidelines. A tailored survey with closed and open questions was used to obtain complementarity data on the topic i.e. to identify the most frequent life situations for children with disabilities for which a product or technology could be useful and drill deeper in these situations with responders' personal experiences to characterize those situations and identify wished solutions.

Survey's development The survey was developed by a group involving three Physical Medicine and Rehabilitation physicians and two occupational therapists. The conceptual framework of the ICF (International Classification of Functioning, Disability and health) which recognizes the role of environmental factors in the creation of disability was used. The survey was pilot tested by two mothers of children with disabilities and an adult who has had a disability since childhood. Comments were considered to improve the survey in a second version.

It was developed using an online tool (google form). Three versions were developed targeting the three participant profiles: persons with childhood onset disabilities, their relatives and the professionals who work with them. Each version was composed of 14 to 16 questions (in 6 pages). Firstly, participants had access to a description of the study with a dedicated picture so that making everyone aware of the project, and precising the general objective of the study. Then, questions were asked on epidemiological data. In a second step, a closed multiple-choice question was presented with a pre-established list of life situations of a regular day. Responders had to select the life situations which they evaluated as the most difficult for children with disabilities to be involved in. Respondents could tick as many items as they wished. All items were extracted from validated scales ("Life H": assesment of Life habits/ "ABILHAND assessment" / "ABILOCO KIDS"/ "PEDI": Paediatric Evaluation of Disability Inventory / "ACTIVLIM-CP"). The list was proposed in a chronological order in order to help the responder think of his own life. Then, open questions invited the respondents to precise the ticked items. The first open question proposed to precisely describe examples from the respondents' own experience (hereinafter referred to as "difficulties") in regular weekdays. Then they had to describe wished strategies that could allow an improvement (hereinafter referred to as "solutions"). Eventually, these last three questions were repeated but dealing with weekend and holidays situations instead of regular weekday situations. The survey was conceived to be short and take less than 10 minutes. Respondents could review and change their answers. No completeness check was proposed. Responders could not be identified from the survey (no identity data, no email or Internet Protocol (IP) address), thus anonymity was guaranteed.

Survey's distribution Participants were surveyed through convenience and snowball sampling to obtain data from participants with a wide range of situations between March and December 2019. The survey was promoted in France through "SFERHE" (Société Francophone d'Etudes et de Recherche sur les Handicaps de l'Enfance) and through the "EACD" (European Academy of Childhood Disability). A leaflet was prepared to present the project. It was posted in hospitals and distributed on social media (Linked in, Facebook, Twitter), and by e-mail. To facilitate the diffusion, the survey was addressed to families and patients' organisations (FFAIMC, "Fondation PC", "AFM"), professional networks ("réseaux maladies rares") and directly promoted during professional events (e.g. "EACD 2019 Paris", "SOFMER 2019 Bordeaux"). Participants answered voluntarily, no incentive was proposed.

ELIGIBILITY:
Inclusion Criteria:

* Persons with disabilities, their families and professionals who work with them

Exclusion Criteria:

1. non-French respondents
2. duplicates
3. void answers

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Three participant profiles are targeted to collect information about life situations during which a technical solution might be useful for children with disabilities: children and young adults with disabilities since childhood, their relatives (family and friendly network) and the professionals who work with them
Sampling Method: Non-Probability Sample
Enrollment: 1055 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Survey- quantitative data | From March 2019 to January 2020
  Quantitative data: identify the frequent difficult life situations for which a technical solution could be useful for children with disabilities
Survey- qualitative data | From March 2019 to January 2020
  Qualitative data: drill deeper in these situations with responders' personal experiences

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Brochard, Study Director — CHRU de Brest, Brest, France; Christelle Pons, Principal Investigator — Fondation Ildys
Locations (1):
- CHRU de Brest, Brest, France